CLINICAL TRIAL: NCT01176396
Title: CAMBRA - PBRN Caries Management By Risk Assessment In A Practice-Based Research Network
Acronym: CAMBRA-PBRN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Dental Association Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCSF A113385
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Dental Caries
Keywords: Dental Caries; Preventive Dentistry; Dental Prophylaxis; Dental Care
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caries prevention active intervention (Active Comparator): Patients receive CAMBRA related products like CHX, 5000ppm F-toothpaste etc according to their risk level
  Interventions: Other: Caries prevention active intervention
- control treatment (Placebo Comparator): Patients receive treatment according to standard of care
  Interventions: Other: control treatment

INTERVENTIONS:
Other: Caries prevention active intervention — Subjects will be treated related to their caries risk:
  "Low Caries Risk"
  The intervention and control treatments for low caries risk are the same:
  4 bitewing radiographs dental prophylaxis Oral Hygiene instruction OTC toothpaste with fluoride (1,100 ppm F) 2x daily Periodic oral exam after 12 months Bitewings after 12 months
  "Moderate Caries Risk" In addition to the treatment above the intervention group receives OTC fluoride rinse as well as xylitol candies or gums.
  "High Caries Risk" The high caries risk level subjects will receive a prescription 5,000 ppm F toothpaste, will rinse 1 day for one week per months with a Chlorhexidine rinse to reduce the bacteria level, and receive a fluoride varnish in the dental office.
  Arms: Caries prevention active intervention
Other: control treatment — Subjects will be treated related to their caries risk:
  "Low Caries Risk"
  The intervention and control treatments for low caries risk are the same:
  4 bitewing radiographs dental prophylaxis (if prescribed) Oral Hygiene instruction OTC toothpaste with fluoride (1,100 ppm F) as currently used by patient Periodic oral exam after 12 months Bitewings after 12 months
  "Moderate Caries Risk" "Control" group receives regular dental care (placebo rinse and gums without active ingredients allow blinding).
  "High Caries Risk" The control treatment group receives regular dental care (regular 1,100 ppm F toothpaste, a placebo rinse without antibacterial ingredients and placebo varnish to allow blinding).
  Arms: control treatment

SUMMARY:
The goal of this project is to create a Practice Based Research Network with 30 researcher dentists calibrated on the administration of a caries risk assessment and the treatment modalities recommended based on the caries risk assessment results (Caries Management by Risk Assessment - CAMBRA), and to conduct a 2-year CAMBRA study in those dental offices. Participating dentists will be a mix of general practitioners and pediatric dentists selected from private practice, part time university faculty, large group practices, or community clinics. Participating practices will collect baseline data and patient progress and report on patient acceptance and compliance, and the effectiveness of treatment.

The program's duration is anticipated to be approximately four years. Year one will be dedicated to program, protocol and evaluation design, and recruitment, selection and calibration of researcher dentists. Years two and three will be the research and data collection time period, and year four will be dedicated to evaluation.

DETAILED DESCRIPTION:
The clinical part of the project will prove that CAMBRA principles can successfully be disseminated into everyday dental practices and that by applying the principles of Caries Management by Risk Assessment to subjects in those practices a major reduction in caries can be seen in the intervention group in comparison to the control group. At the end of the two year clinical part performed in the Practice Based Research Network data will show that the positive results of the first CAMBRA study achieved in the university setting at UCSF can also be accomplished in a dental practice setting to the benefit of patients. If CAMBRA can be successfully disseminated into dental practices dental care costs can significantly be reduced.

The overall study objective is to build a Practice Based Research Network (PBRN) and to conduct in this setting a 2-year randomized, controlled, double blind clinical trial to provide clinical evidence that scientifically based caries risk assessment, in conjunction with aggressive preventive measures and conservative restorations will result in dramatically reduced further caries increment. If successful this study performed in a PBRN will provide substantial evidence for changing the practice of caries management. The planned study is a double blind practice-based clinical study. The California Dental Association Foundation will help to select up to 30 participating dentists. Practitioners will perform a Caries Management by Risk Assessment (CAMBRA) evaluation and will instruct and provide treatment suggestions for the study subjects according to the CAMBRA protocol.

The hypothesis to be tested is that caries management based on caries-risk status (low, moderate or high) will significantly reduce the need for caries restorative treatment over two (plus) years compared to usual dental treatment in the practice based setting. The primary outcome measure will be caries increment.

At the end of the two year clinical part performed in the Practice Based Research Network data will show that the positive results of the first CAMBRA study achieved in the university setting at UCSF can also be accomplished in a dental practice setting to the benefit of patients. If CAMBRA can be successfully implemented into dental practices in the future dental care costs can significantly be reduced.

ELIGIBILITY:
Inclusion Criteria:

* These criteria will not be based on race or gender.
* Participants will be new patients and must:
* be at least 12 years old and not older than 65 years
* be able to give informed consent in English
* be unlikely to move from the area during the study period (as determined by residential history and questioning, and be unlikely to move in the next 2.5 years for work, educational, or personal reasons.)
* be willing to participate regardless of group assignment
* be willing to comply with all study procedures and protocol
* be dentate with at least sixteen teeth
* will have all treatment needs for caries completed within three months of entry into the study

Exclusion Criteria:

* People who want to limit radiation exposure from dental radiographs
* Persons with:
* significant past or current medical problem history especially conditions that may affect oral health or oral flora (i.e., diabetes, HIV, heart conditions that require antibiotic prophylaxis)
* medication use that may affect the oral flora or salivary flow (e.g., antibiotic use in the past three months, drugs associated with dry mouth/xerostomia)
* root caries at enrollment (study will focus on coronal caries)
* periodontal disease that requires surgery, chemotherapeutic agents, or frequent prophys
* another household member participating in the study (to prevent sharing F, CHX rinses, etc.)
* drug or alcohol addiction, or other conditions that may decrease the likelihood of adhering to study protocol
* missed screening visit without cancellation or rescheduling
* rescheduled screening visit more than once
* subjects with extreme high caries risk
* sensitive to Chlorhexidine or the ethyl alcohol vehicle in CHX

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
caries increment | 2 years

SECONDARY OUTCOMES:
changes in mutans streptococci (MS), and lactobacilli (LB) in whole saliva | 2 years
change in caries risk category over time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rechmann, DDS, PhD, Principal Investigator — University of California, San Francisco, School of Dentistry; John DB Featherstone, MSc, PhD, Principal Investigator — University of California, San Francisco, School of Dentistry
Locations (1):
- UCSF School of Dentistry - Dental Offices in Bay Area, San Francisco, California, United States

REFERENCES:
- [Background] Kaste LM, Selwitz RH, Oldakowski RJ, Brunelle JA, Winn DM, Brown LJ. Coronal caries in the primary and permanent dentition of children and adolescents 1-17 years of age: United States, 1988-1991. J Dent Res. 1996 Feb;75 Spec No:631-41. doi: 10.1177/002203459607502S03. PMID 8594087
- [Background] NCHS. National Center for Heath Statistics, Government Printing Office, Washington D.C. 1974.
- [Background] NIDR. The prevalence of dental caries in United States children: The National Dental Caries Prevalence Survey: 1979-80. NIH Publication No. 82-2245. National Institutes of Health 1981.
- [Background] Brunelle JA. Oral Health of United States Children: The National Survey of Dental caries in US School Children:1986-87. National Institute of Dental Research 1989.
- [Background] Speechley M, Johnston DW. Some evidence from Ontario, Canada, of a reversal in the dental caries decline. Caries Res. 1996;30(6):423-7. doi: 10.1159/000262354. PMID 8946102
- [Background] Beltran-Aguilar ED, Barker LK, Canto MT, Dye BA, Gooch BF, Griffin SO, Hyman J, Jaramillo F, Kingman A, Nowjack-Raymer R, Selwitz RH, Wu T; Centers for Disease Control and Prevention (CDC). Surveillance for dental caries, dental sealants, tooth retention, edentulism, and enamel fluorosis--United States, 1988-1994 and 1999-2002. MMWR Surveill Summ. 2005 Aug 26;54(3):1-43. PMID 16121123
- [Background] Bowen WH. Do we need to be concerned about dental caries in the coming millennium? Crit Rev Oral Biol Med. 2002;13(2):126-31. doi: 10.1177/154411130201300203. PMID 12097355
- [Background] Ismail AI, Burt BA, Brunelle JA. Prevalence of total tooth loss, dental caries, and periodontal disease in Mexican-American adults: results from the southwestern HHANES. J Dent Res. 1987 Jun;66(6):1183-8. doi: 10.1177/00220345870660061801. PMID 3476591
- [Background] Ismail AL, Burt BA, Brunelle JA. Prevalence of dental caries and periodontal disease in Mexican American children aged 5 to 17 years: results from southwestern HHANES, 1982-83. National Health and Nutrition Examination Survey. Am J Public Health. 1987 Aug;77(8):967-70. doi: 10.2105/ajph.77.8.967. PMID 3605476
- [Background] Featherstone JDB, Gansky SA, Hoover CI, Rapozo-Hilo ML, Weintraub JA, White JM, et al. Chlorehexidine and fluoride therapy reduces caries risk. J Dent Res 2005;84 [Spec Iss A, abstract 0023].
- [Background] Hoover CI, Weintraub JA, Gansky SA, White JM, Wilson RS, Featherstone JDB. Effect of a caries management regimen on cariogenic bacterial population. J Dent Res. 2004;83 [Spec Iss A, abstract 0779].
- [Background] Hoover CI, Weintraub JA, Gansky SA, White JM, Wilson JA, Featherstone JDB. Effect of restorations and Bacterial Challenge Management on Cariogenic Bacteria. J Dent Res. 2005;84 [Spec Iss A, abstract 3254].
- [Background] Domejean-Orliaguet S, Gansky SA, Featherstone JD. Caries risk assessment in an educational environment. J Dent Educ. 2006 Dec;70(12):1346-54. PMID 17170326
- [Background] Young DA, Featherstone JD, Roth JR, Anderson M, Autio-Gold J, Christensen GJ, Fontana M, Kutsch VK, Peters MC, Simonsen RJ, Wolff MS. Caries management by risk assessment: implementation guidelines. J Calif Dent Assoc. 2007 Nov;35(11):799-805. PMID 18080486
- [Background] Young DA, Featherstone JD, Roth JR. Curing the silent epidemic: caries management in the 21st century and beyond. J Calif Dent Assoc. 2007 Oct;35(10):681-5. PMID 18044376
- [Background] Featherstone JD, Domejean-Orliaguet S, Jenson L, Wolff M, Young DA. Caries risk assessment in practice for age 6 through adult. J Calif Dent Assoc. 2007 Oct;35(10):703-7, 710-3. PMID 18044378
- [Background] American Dental Association. Fluoridation Facts. Chicago. IL; 2005.
- [Background] Institute of Medicine, Food and Nutrition Board. Dietary reference intakes for calcium, phosphorus, magnesium, vitamin D and fluoride. Report of the Standing Committee on the Scientific Evaluation of Dietary Reference Intakes. Washington, DC: National Academy Press; 1997.
- [Background] Hodge HC. The safety of fluoride tablets or drops. In: Johansen E, Tavaes DR, Olsen TO, editors. Continuing evaluation of the use of fluorides. Bolder, CO: Westview Press; 1979. p. 253-75.
- [Background] Milgrom P, Ly KA, Roberts MC, Rothen M, Mueller G, Yamaguchi DK. Mutans streptococci dose response to xylitol chewing gum. J Dent Res. 2006 Feb;85(2):177-81. doi: 10.1177/154405910608500212. PMID 16434738
- [Background] Milgrom P, Ly KA, Tut OK, Mancl L, Roberts MC, Briand K, Gancio MJ. Xylitol pediatric topical oral syrup to prevent dental caries: a double-blind randomized clinical trial of efficacy. Arch Pediatr Adolesc Med. 2009 Jul;163(7):601-7. doi: 10.1001/archpediatrics.2009.77. PMID 19581542
- [Background] Vernacchio L, Vezina RM, Mitchell AA. Tolerability of oral xylitol solution in young children: implications for otitis media prophylaxis. Int J Pediatr Otorhinolaryngol. 2007 Jan;71(1):89-94. doi: 10.1016/j.ijporl.2006.09.008. Epub 2006 Nov 9. PMID 17097152
- [Background] Oku T, Nakamura S. Threshold for transitory diarrhea induced by ingestion of xylitol and lactitol in young male and female adults. J Nutr Sci Vitaminol (Tokyo). 2007 Feb;53(1):13-20. doi: 10.3177/jnsv.53.13. PMID 17484374
- [Derived] Rechmann P, Chaffee BW, Rechmann BMT, Featherstone JDB. Changes in Caries Risk in a Practice-Based Randomized Controlled Trial. Adv Dent Res. 2018 Feb;29(1):15-23. doi: 10.1177/0022034517737022. PMID 29355409